CLINICAL TRIAL: NCT04868942
Title: Protective Measures Against SARS-CoV-2 Contamination of Healthy Voluntary Young Students During a Concert of Actual Music
Brief Title: Protective Measures Against SARS-CoV-2 Contamination of Young Healthy Volunteers During a Concert of Actual Music
Acronym: CONCERTSAFE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study didn't get the authorization from health authority
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Sciences Economiques et Sociales de la Santé & Traitement de l'Information Médicale (Unknown); Faculté des Sciences Médicales et Paramédicales (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ANRS0004s
Record Dates: First submitted 2021-04-16; First posted 2021-05-03 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Corona Virus Infection
Keywords: Coronavirus; Healthy volunteers; Social distancing; Prevention; Face masks
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: A randomised, monocentric, open-label, non-inferiority study comparing, in two phases, a group of volunteers participating in a concert, protected by established protection measures (protection kit, distancing, flow management, health mediation), to a group with no other constraints than national recommendations and obligations (2 concerts, one control group at each concert).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participant assisting to the event (Experimental): Attending to musical event protected by established protection measures (protection kit, distancing, flow management, health mediation).
  Interventions: Other: Assisting to the event
- Participant with no other constraints than national recommendations (No Intervention): A group control participant will not attend to the event

INTERVENTIONS:
Other: Assisting to the event — Participant will attend a concert respecting the Following measures :
  * Individual protection kit: disposable FFP2 masks (3), Hydroalcoholic solution, disposable tissues, garbage bag, water bottle
  * Health mediation, information on barrier measures
  * Physical distancing (sitting participation)
  * Person flow management
  Other Names: Attend a concert
  Arms: Participant assisting to the event

SUMMARY:
The aim of this study is to assess whether the protective measures can limit the contaminations by SARS-CoV-2 during the participation in a concert at a non-inferior level to a non-concert / current life situation. A randomized, monocentric, open-label, non-inferiority study comparing, in two phases, a group of volunteers participating in a concert, protected by established protection measures, to a group with no other constraints than national recommendations and obligations (2 concerts, one control group at each concert). Volunteer students, between 18 and 30 years old, at Aix-Marseille University, will be recruited.

DETAILED DESCRIPTION:
Objectives

Primary objective To assess whether the protective measures implemented (individual protection kit including disposable FFP2 (filtering facepiece) masks, hydro-alcoholic solution, water bottle, disposable tissues, waste bag, physical distancing, flow management and health mediation) make it possible to limit contamination by SARS-CoV-2 during participation in a concert (lasting 2 hours) at a non-inferior level to a non-concert situation

Secondary objectives

* To assess whether the protective measures implemented (individual protection kit including disposable FFP2 masks, hydro-alcoholic solution, water bottle, disposable tissues, waste bag, physical distancing, flow management and health mediation) make it possible to limit contamination by other circulating respiratory viruses during participation in a concert (lasting 2 hours) at a non-inferior level to a non-concert situation
* To assess whether the protection against viral contamination in the absence of a one-seat gap between 2 volunteers is non-inferior to the protection induced by one-seat gap (sub-group of volunteers)
* To assess knowledge, attitudes and practices regarding COVID-19
* To assess the level of compliance and adherence to the prevention measures implemented during the concert
* To assess SARS-CoV-2 serology prevalence in volunteers
* To identify SARS-CoV-2 variants by sequencing SARS-CoV-2 PCR positive cases

Methodology / design A randomized, monocentric, open-label, non-inferiority study comparing, in two phases, a group of volunteers participating in a concert, protected by established protection measures (protection kit, distancing, flow management, health mediation), to a group with no other constraints than national recommendations and obligations (2 concerts, one control group at each concert).

Sample size

4500 participants, in 2 phases: Phase A: Concert A group, n=1125; Control A group, n=1125 Phase B (15 days later): Concert B group, n=1125; Control B group, n=1125

Endpoints

Primary Endpoint:

Conversion of salivary SARS-CoV-2 carriage detected by molecular biology at Day 6 or 7 after each event

Secondary endpoints:

* Conversion of salivary carriage of other respiratory viruses detected by molecular biology at Day 6 or 7 after each event
* Level of knowledge about COVID-19 and methods of protection
* Verbatim from the qualitative interview on knowledge, attitudes and practices
* Adherence score for protective measures
* Percentage of initially positive SARS-CoV-2 serology in the volunteer sample
* Percentages of SARS-CoV-2 variants among positive samples (for each variant)

Intervention

During the music concert (2 hours), prevention measures:

* Individual protection kit: disposable FFP2 masks (3), hydro-alcoholic solution, disposable tissues, garbage bag, water bottle
* Health mediation, information on barrier measures
* Physical distancing (sitting participation)
* Person flow management

Statistical Plan

Primary analysis:

The intervention effect will be estimated by the difference in SARS-CoV-2 conversion rates (PCR).

The main non-inferiority analysis will be performed by interval estimation of the difference in PCR SARS-CoV-2 conversion rates, in Per Protocol (each volunteer being associated with the concert or control group according to his or her actual participation), over the 2 concerts (using a multilevel mixed model, with random period effect). An Intention-to-Treat analysis will also be performed.

Secondary analyses:

* Analysis of individual knowledge and behavior, and adherence to protection measures (Q1- questionnaire Q1, Q2 and Q3): unsupervised exploratory analyses - classification on principal component analysis
* Estimation of the difference in PCR conversion rates (SARS-CoV-2 and other respiratory viruses) adjusted for the level of knowledge and behavior obtained from the questionnaires, for the collective level of protection observed during the concert (ad hoc observations), and for the epidemic situation at the time of the concerts. Estimations will be provided by using a multilevel multivariate logistic model. This approach will eventually allow us to introduce a random period effect to consider the temporality of the measurements. Finally, we analyze the level of the epidemic by IRIS (smallest french geographical area) each week, in collaboration with the ARS-PACA (Health Regional Agency - Agence Regionale de Santé - Provence Alpes Cote d'Azur) and SPF (French National Public Health Agency - Santé Publique France). If necessary, an adjustment on this possible spatial effect will be made, based on the address of the volunteers, to estimate the risk of contamination of the control group (exponential-power variogram)
* Serology prevalence will be estimated, and associated behavioral factors will be assessed by using multilevel multivariate logistic regression
* Analyses will be performed in Per Protocol and Intent to Treat
* A secondary analysis with imputation of missing data will be performed as a sensitivity analysis (after testing the hypothesis of missing at random)

A 5% significance level will be used for decision making, but the probabilities will be interpreted accordingly.

Provisional timetable: follow-up of volunteers

D-30 to D-16: logistic organization D-15: information about the study, communication in the media, call for volunteers D-10 to D-2: selection of eligible volunteers

Phase A (n=2250) D-2 to D-1: Phase A Inclusion visit (medical verification of inclusion criteria, information leaflet, consent form), 1:1 randomization into two groups of 1125 volunteers (Concert A and Control A); self-collection of PS-A1 saliva sample ("Prélèvement Salivaire") and Q-A1-baseline questionnaire at one of the dedicated university campuses, explanation of instructions; self-collection for serology D0: Concert A group (n=1125) participating to the first concert after receiving the health kit and instructions at the entrance vs Controls A (n=1125), "usual" life D1 to D2: Q-A2 adherence questionnaire D6 to D7: Phase A control visit; self-collection of the PS-A2 saliva sample at one of the dedicated university campuses, reminder of instructions; interviews (focus group n=10) for a sub-group of volunteers.

D0 to D10: Medical follow-up of Phase A volunteers; Q-A3 follow-up questionnaire

Phase B (n=2250) D13 to D14: Phase B Inclusion visit (medical verification of inclusion criteria, information leaflet, consent form), 1:1 randomization into two groups of 1125 volunteers (Concert B and Control B); self-collection of PS-B1 saliva sample and Q-B1-baseline questionnaire at one of the dedicated university campuses, explanation of instructions; self-collection for serology D15: Concert B group (n=1125) participating to the first concert after receiving the health kit and instructions at the entrance vs Controls B (n=1125), "usual" life D16 to D17: Q-B2 adherence questionnaire D21 to D22: Phase B control visit; self-collection of the PS-B2 saliva sample at one of the dedicated university campuses, reminder of instructions; interviews (focus group n=10) for a sub-group of volunteers.

D14 to D25: Medical follow-up of Phase B volunteers; Q-B3 follow-up questionnaire

Analyses

D10 to D32: Biological sample processing D25 to D40: Questionnaire processing D35 to D65: Primary statistical analyses D65-D365: Secondary analyses

ELIGIBILITY:
Inclusion Criteria:

* Student at Aix Marseille University
* who has declared that he or she does not carry any risk factor for severe forms of the disease (HCSP criteria of 29/10/2020)
* who has declared that he or she does not live under the same roof as a person who does carry such factors, and committed to strictly following the study's health protocol,
* carrying a smartphone which is registered on the "TousAntiCovid" application (with Bluetooth activation), and agreeing to install the Maela application on the smartphone for remote medical monitoring.

Exclusion Criteria:

* Volunteer with clinical signs of acute respiratory infectious disease
* Volunteer living with a person with clinical signs of acute respiratory infectious disease
* Volunteer with a risk factor for severe COVID-19
* Volunteer who had a COVID-19 infection in the 3 months prior to the study
* Volunteer who are not affiliated to the social security system
* Volunteer vaccinated against COVID-19
* Pregnant women and people living with pregnant women
* Persons deprived of liberty
* Adult with legal protection
* Volunteer unable to comply with protective measures, at the concert or at home
* Volunteer participating in another clinical research study

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 conversion rates | 6 to 7 days after attending to the musical event
  PCR on saliva sample

SECONDARY OUTCOMES:
Respiratory virus conversion rates | 6 to 7 days after attending the concert
  PCR on saliva sample
Types and importance of barriers to prevention measures | 1 to 2 day before attending the concert
  Participant satisfaction survey using context-specific measures. A-Measures of perceived discomfort and perceived degradation of feelings Five points qualitative bipolar likert scale (four preventive behaviours items) minimum -2 to maximum 2, higher scores mean a better outcome.
  1. use of face mask
  2. physical distancing
  3. screening before admission
  4. motion monitoring in the concert hall
  B-Measure of social gathering behaviors Five points qualitative bipolar likert scale (four behavioural items) minimum -2 to maximum 2, higher scores mean a better outcome.
  1. Socializing: talking to people
  2. Socializing: meeting new people
  3. Showing pleasure: singing or shouting
  4. Showing pleasure: Dancing
  C-Measures overall satisfaction, using a single numeric item scale rated from 0 to 10 and an adapted Net Promoter Score scale.
  Higher scores mean a better outcome.
Types and importance of levers for adherence to prevention measures | 1 to 2 days after attending the concert
  Focus groups (after the concert)
Seroprevalence of SARS-CoV-2 in volunteers | 1 to 2 days before attending the concert
  Assess SARS-CoV-2 seroprevalence in volunteers
SARS-CoV-2 variants among participant positive cases | 6 to 7 days after attending the concert
  Identify SARS-CoV-2 variants by sequencing SARS-CoV-2 PCR positive cases

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Simon, Prof, Principal Investigator — Faculté des Sciences Médicales et Paramédicales

IPD SHARING:
Plan to Share IPD: No